CLINICAL TRIAL: NCT06154577
Title: Tongue Morphology and Posterior Airway Space as Predictors of Response in Patientswith Hypoglossal Nerve Stimulation Therapy
Status: Completed | Type: Observational
Sponsor: Cantonal Hosptal, Baselland (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-00117
Record Dates: First submitted 2023-11-16; First posted 2023-12-04 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Obstructive Sleep Apnea; Sleep-Disordered Breathing
Keywords: hypoglossal nerve stimulation; ultrasonography
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obstructive sleep apnea patients: 39 obstructive sleep apnea patients with hypoglossal nerve stimulation
  Interventions: Diagnostic Test: Ultrasonography
- Healthy controls: 15 healthy control participants
  Interventions: Diagnostic Test: Ultrasonography

INTERVENTIONS:
Diagnostic Test: Ultrasonography — Assessment of tongue morphology and posterior airway space using ultrasonography (AmCAD-UO, CE mark NB1639)

SUMMARY:
Hypoglossal nerve stimulation (HNS) plays an increasingly important role in managing patients with obstructive sleep apnea (OSA) who do not tolerate CPAP therapy and are not eligible for other alternative treatment options, such as mandibular advancement devices or positional therapy. The posterior upper airway space dimensions are crucial in managing patients with HNS in the patient selection process and therapy control. The lateral collapse of the upper airway is of crucial importance. Lateral collapse at the palatal level and of the oropharyngeal walls is a well-established negative predictive factor for therapeutic success. Patients with complete concentric collapse at the palatal level (pCCC) in drug-induced sedation endoscopy (DISE) must be excluded from the implantation of HNS, which is cumbersome and invasive. Endoscopy has the inherent limitation that only one level can be observed at a given time, and assessment is possibly hampered by phlegm.

During activation and titration of HNS, tongue protrusion is observed in the awake patient. However, this method does not allow for assessing the opening of the retroglossal (RG) and retropalatal (RP) airway space, which is the ultimate therapeutic goal. Insufficient opening of the airway is the reason for non-responders with HNS. Insufficient upper airway opening can be either at the retropalatal or retroglossal level. The study aims to identify insufficient airway openings better using sub-mental ultrasonography. Sub-mental standardized and orientated ultrasonography offers a quantitative, reproducible way of assessing transverse upper airway dimensions and anatomic features of the upper airway in a rapid and non-invasive manner. In addition, anatomic characteristics of the airway's adjacent tissue, such as the size and shape of the tongue, may also have an impact on the effectiveness of HNS. Tongue morphology and posterior airway space assessment could be used in preoperative evaluation and during therapeutic titration of HNS. The clinical routine could be included tongue morphology and posterior airway space assessment without additional patient risks. However, the clinical value of assessing posterior airway space and tongue morphology in patients with HNS is yet unknown.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 year
* patients with a hypoglossal nerve implantation
* control group: 15 subjects without OSA (AHI<10/h)
* written informed consent
* sufficient knowledge of German or French to understand informed consent

Exclusion Criteria:

* Patients younger than 18 years
* unwillingness to give informed consent
* incapable of performing Müller's maneuver
* history of head and neck surgery other than HNS, tonsillectomy, and maxillomandibular advancement
* diagnosis of congestive heart failure or chronic pulmonary disease
* diagnosis of co-morbid sleep disorders, including central sleep apnea
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 39 obstructive sleep apnea patients with hypoglossal nerve stimulation and 15 subjects in the control group
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Prediction of therapeutic success with hypoglossal nerve stimulation | Most recent sleep testing before examination after HNS implantation, a maximum of 6 months before examination
  Success is defined as apnea-hypopnea index in the most recent sleep testing ≤ 20/h and 50% reduction from baseline

SECONDARY OUTCOMES:
Prediction of AHI reduction, defined as the difference between pre- and postoperative AHI, with HNS based on tongue morphology and posterior airway space. | Most recent sleep testing before examination after HNS implantation, a maximum of 6 months before examination
  AHI reduction is defined as apnea-hypopnea index in the most recent sleep compared to the baseline value before HNS implantation
Comparison of pharyngeal dimensions between visual assessment and tongue morphology and posterior airway space | through study completion, from 15.05.2023 to 14.05.2024
  Visual assessment is performed both by DISE and wake transnasal endoscopy. Tongue morphology and posterior airway space is analyzed using ultrasonography
Therapeutical guidance using tongue morphology and posterior airway space to identify the obstructing upper airway segment compared to wake fiberoptic endoscopy during HGS in non-responders. | through study completion, from 15.05.2023 to 14.05.2024
  Changes to therapeutic HNS settings during study visit
Patient comfort rated by the patients for wake transnasal endoscopy and sub-mental ultrasonography | through study completion, from 15.05.2023 to 14.05.2024
  Rated on a visual analog scale (VAS) from 0 to 10 (0 meaning no discomfort; 10 meaning very uncomfortable
Information gain through from tongue morphology and posterior airway space imaging | through study completion, from 15.05.2023 to 14.05.2024
  Rating by the physician if the additional information gained from tongue morphology and posterior airway space imaging at functional stimulation threshold is a valuable adjunct to the oral observation of tongue protrusion rated on a VAS
Comparison of pharyngeal dimensions of healthy and patients with OSA and HNS | through study completion, from 15.05.2023 to 14.05.2024
  Pharyngeal dimensions measured using ultrasonography

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Kantonsspital Baselland, Liestal, Basel-Landschaft
  - University Hospital Bern, Inselspital, Bern

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tschopp S, Janjic V, Lee Y, Chen A, Chao PY, Caversaccio M, Borner U, Tschopp K. Backscattered Ultrasonographic Imaging of the Tongue and Outcome in Hypoglossal Nerve Stimulation. Otolaryngol Head Neck Surg. 2025 Jun;172(6):2134-2140. doi: 10.1002/ohn.1251. Epub 2025 Apr 7. PMID 40192006